CLINICAL TRIAL: NCT06621745
Title: A Mobile Application-based Gratitude Intervention's Psychological Effects
Brief Title: A Gratitude Intervention App to Reduce Symptoms of Depression, Anxiety and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canada Foundation for Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-5460_GIA
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Depression; Anxiety; Stress
Keywords: Gratitude intervention; Smartphone app; Gratitude exercises; Psychological well-being; Student mental health
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study used a randomized experimental design to test the effectiveness of a gratitude intervention smartphone app. Participants were asked to answer 90 questions in an online survey on emotional well-being and personality traits at the beginning and end of the three-week research period. The intervention group used the Gratitude Intervention App (GIA), and the Predicting Risk and Outcomes of Social InTerActions (PROSIT) app, which is a mobile sensing app. All participants used the PROSIT app in the background of their mobile devices throughout the three-week study period. In addition, those allocated to the intervention group practiced gratitude intervention tasks during the same three-week period using the GIA app. This study was approved by the Dalhousie University Research Ethics Board (REB 2021-5460).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gratitude Intervention Group (Experimental): The intervention group used the Gratitude Intervention App (GIA), and the Predicting Risk and Outcomes of Social InTerActions (PROSIT) app, which is a mobile sensing app.
  Interventions: Behavioral: Gratitude Intervention App
- Control Non-gratitude Intervention Group (No Intervention): Participants in the control group downloaded and used only the PROSIT app, they did not use the Gratitude Intervention App (GIA).

INTERVENTIONS:
Behavioral: Gratitude Intervention App — The GIA app, an iOS application designed for this study, is based on effective gratitude interventions and tailored for youth. Access required a unique login. It features five exercises: a journal, photo book, imagine exercise, speech exercise, and meditation. The journal encourages daily entries. The photo book involves uploading photos of things users are grateful for, promoting mindfulness. The imagine exercise reflects on gratitude, while the speech exercise records users' gratitude. The meditation exercise enhances well-being. During the three-week study, daily notifications prompted exercise completion. The app, green and white with a flower-heart icon, offers email support for technical issues.
  Other Names: GIA
  Arms: Gratitude Intervention Group

SUMMARY:
The goal of this clinical trial is to examine whether a newly developed gratitude intervention app can effectively improve psychological functioning, as measured by depression, anxiety, and stress symptoms, positive and negative affect

The main questions it aims to answer are:

1. Will people who are in the intervention group feel more positive emotions and experience fewer negative emotions such as stress, anxiety, and depression after three weeks?

Researchers will compare the intervention to a control group (a group not given the gratitude intervention) to see if the intervention works to improve psychological functioning.

Participants will:

* Complete an online survey on emotional well-being and personality traits at the beginning and end of the three-week study, with daily mood ratings and stress assessments every three days.
* Participants in the intervention group will use a mobile app to practice gratitude exercises.

DETAILED DESCRIPTION:
Background: Gratitude interventions have been shown to decrease depression, stress and anxiety symptoms, support enhanced coping with health-related problems and might improve both psychological and physical functioning in areas. However, results have been mixed with effects varying by outcome, duration, follow-up length, format, and age. A recent meta-analysis including 27 studies focusing more specifically on symptoms of depression and anxiety suggest there is a limited effect of gratitude interventions on reducing symptoms of depression and anxiety at post-intervention and follow-up.

Objective: Thus, the present study aims to implement a three-week gratitude intervention including five different types of gratitude tasks embedded in a mobile sensing application and examine the intervention's psychological effects.

Method: Participants will be recruited and randomly allocated into the intervention and the control group. The study will measure depression, anxiety and stress symptoms, positive and negative affect, negative affectivity and social inhibition before and after the three-week intervention period as psychological variables. It will analyze the effect of the gratitude intervention on the measured variables as well as examine the impact of negative affectivity and social inhibition on depression, anxiety and stress symptoms.

Implications: If the intervention is shown to effectively reduce psychological problems, it will be tested and implemented to support the well-being of university students as a stand-alone tool.

The study will examine whether the gratitude intervention can effectively reduce depression, anxiety and stress symptoms. We intend to recruit 120 participants. Extending previous research, it will also examine whether negative affectivity and social inhibition have an impact on the measured outcomes and whether the intervention can influence these traits.

It is hypothesized that:

1. Positive affect will increase, while negative affect, stress, anxiety and depression symptoms will decrease from before to after the three weeks in the group that practices the gratitude intervention tasks (intervention group) compared to the group which doesn't (control group).
2. Negative affectivity and social inhibition will decrease from before to after the three weeks in the intervention group in comparison to the control group.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 18-30, with access to an iPhone, and English speaking.

Exclusion Criteria:

* any self-reported cardiovascular disease; endocrine disease, kidney disease, tumor, hypertension, coarctation of the aorta, fibromuscular dysplasia, sleep apnea, which can impact the function of the cardiovascular system, as well as any current mental health treatment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Depression, anxiety, and stress | three weeks
  Participant's depression, anxiety, and stress levels were measured with the Depression, Anxiety, and Stress Scale (DASS-21), which is a set of three self-report scales each consisting of seven items to measure the individual's emotional states of depression ("I couldn't seem to experience any positive feeling at all"), anxiety ("I felt I was close to panic"), and stress ("I found it difficult to relax"). Participants rated how much each statement applied to them in the past week, from 0 ("Did not apply to me at all") to 3 ("Applied to me very much or most of the time"). High scores indicate higher levels of symptoms of anxiety, depression, and stress. There are subscale score cut-offs for normal, mild, moderate, severe, and extremely severe emotional states. Participants were considered to show at least moderate symptomatology if they scored higher than 7 on the depression subscale, 6 on the anxiety subscale, and 10 on the stress subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Meier, PhD, Principal Investigator — Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Participant data will be made available upon reasonable request to Dr. Sandra Meier (PI).